CLINICAL TRIAL: NCT02506504
Title: Prevention of Post-exercise Muscle Fatigue Using a Non Invasive Ventilation and Effect on Exercise Training in Severe Patients With COPD. QUADRIVEND Study
Brief Title: Prevention of Post-exercise Muscle Fatigue and Effect on Exercise Training in Severe Patients With COPD.
Acronym: QUADRIVEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1308189; 2014-A00145-42 (Other: ANSM)
Record Dates: First submitted 2015-07-16; First posted 2015-07-23 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Lung Diseases
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory help then sham ventilation (Experimental): The initial evaluation is performed using an Inspiratory Pressure Support. After the training, the final evaluation is performed using an Inspiratory help (sham ventilation).
  Interventions: Device: Inspiratory help then sham ventilation
- Sham ventilation then Inspiratory help (Experimental): The initial evaluation is performed using an inspiratory help (sham ventilation).
  After the training, the final evaluation is performed using an Inspiratory Pressure Support.
  Interventions: Device: Sham ventilation then Inspiratory help

INTERVENTIONS:
Device: Inspiratory help then sham ventilation — The Inspiratory Pressure Support is used to increase the intensity and the duration of training session. For the sham ventilation, the device deliver a non effective quantity of oxygen.
  Arms: Inspiratory help then sham ventilation
Device: Sham ventilation then Inspiratory help — The Inspiratory Pressure Support is used to increase the intensity and the duration of training session. For the sham ventilation, the device deliver a non effective quantity of oxygen.
  Arms: Sham ventilation then Inspiratory help

SUMMARY:
In patients with severe Chronic Obstructive Pulmonary Disease (COPD), exercise tolerance is severely impaired due to a ventilatory limitation, levelling off the intensity of exercise. This reduces the physiological benefit of pulmonary rehabilitation. In these patients, it is then proposed to add an Inspiratory Pressure Support (IPS) in order to increase the intensity and the duration of every training session. In a preliminary study, the investigators showed that IPS applied during an exhaustive cycling exercise allowed to prevent the onset of post-exercise quadriceps fatigue evaluated by the endurance time to isotonic quadriceps contractions (TlimQ).

The aim of this study is to determine the relationship between the prevention of post-exercise fatigue (TlimQ) and the change in training load (intensity x time x number of sessions) during a pulmonary rehabilitation programme. At the beginning of the training programme, 25 patients will be evaluated for TlimQ after a cycling exercise (70% maximal workload) with and without IPS in random order. The training load was then monitored at every exercise session of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD patients in stable condition (Gold class 3 or 4)
* Ventilatory limitation to exercise during the incremental cardiopulmonary exercise test (at least one of the following criteria) :
* No breathing reserve
* Exercise hypoventilation (increase arterial PCO2> 5 mmHg)
* Maximal workload <50 Watts

Exclusion Criteria:

* IPS not tolerated during a preliminary cycling exercise test
* Enable to perform the exercise tests or the rehabilitation programme
* Decline to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06-25; Primary Completion 2018-10-22 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Strength of the correlation between the change of TlimQ (min) and the training load calculated as intensity (in watts) x duration of the session (minute) x number of sessions | Visit 24 (week 8)
  At the beginning of the programme, we evaluate the influence of IPS on TlimQ (visits 2 and 3). After the training period, we repeated the same evaluations (visits 23 and 24). Then, we will compare this difference before and after the training period, and we will seek for a relation with the training load.

SECONDARY OUTCOMES:
variation TlimQ of post-exercise without and with IPS | Visit 3 (week 1)
  We compare the endurance time to isotonic quadriceps contractions after a cycling exercice until exhaustion with and without IPS, at the beginning of the training period.
relationship between the change in the endurance to cycling exercise without and with IPS and the change in TlimQ | Visit 24 (week 8)
  we will compare the difference in endurance to exercise with IPS and the difference in endurance to isotonic quadriceps contractions
relationship between the change in the endurance to cycling exercise with IPS and the change in TlimQ | Visit 24 (week 8)
  we will seek for a relationship between the changes in the endurance time to cycling exercise without or with IPS and the variation in endurance to isotonic quadriceps contractions following cycling exercise
variation of TlimQ after a cycling exercice untill fatigue without IPS at the beginning and the end of pulmonary rehabilitation evaluated by the endurance time to isotonic quadriceps contractions | Visit 24 (week 8)
variation of TlimQ after a cycling exercice untill fatigue with IPS at the beginning and the end of pulmonary rehabilitation evaluated by the endurance time to isotonic quadriceps contractions | Visit 24 (week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARTHELEMY, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Clinique Cardio-pneumologique de Durtol, Durtol
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No